CLINICAL TRIAL: NCT02311387
Title: Study of the Seroprevalence and the Incidence of Lassa Fever in the Rural Commune of Sibirila, District of Bougouni, Mali
Brief Title: Seroprevalence and Incidence of Lassa Fever in the Rural Commune of Sibirila, District of Bougouni, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915023; 15-I-N023
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-10-22

CONDITIONS: Lassa Virus Infection
Keywords: Incidence; Prevalence; Human; Mastomys; Serosurvey
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Lassa fever is very similar to other diseases that cause fever, such as malaria and yellow fever. People get Lassa fever from mice. A person can get Lassa fever from mice urine and droppings. When a group of researchers tested the mice in Soromba, Mali, they found that many were infected with Lassa fever. Lassa fever may also be passed through body fluids (like blood or semen) of people infected with Lassa fever. Researchers want to study this disease to help the government better protect the health of people in Sibirila.

Objectives:

- To find out how many people in Sibirila have ever had Lassa fever. Also, to measure how many people get the disease every year.

Eligibility:

- People age 6 months and older who are residents of Soromba, Bamba, or Banzana with no plans to relocate within 1 year.

Design:

* Households will be randomly selected to participate in the study.
* Participants will have up to 20 drops of blood collected from the finger or heel.
* Participants will be asked about their age. They will be asked if they have ever had a fever and if they have ever seen mice in or around their home.
* Researchers will come back in 1 year and take another drop of blood from the participant. Participants will be asked the same questions.
* If a participant has a fever at any time during the year, he or she should go to the health center. Researchers

will collect a few drops of blood to test for Lassa fever.

...

DETAILED DESCRIPTION:
Throughout West Africa as many as 300,000 people are infected annually with Lassa virus, resulting in approximately 5,000 deaths. Most commonly, contact with infected rodent hosts (Mastomys natalensis), or ingestion / inhalation of virus laden particles is the source of human infection. However, person-to-person transmission is also well documented and can result in outbreaks, especially in nosocomial settings. Infection in pregnancy, especially the third trimester, is particularly severe with maternal mortality rates estimated at 20% and fetal mortality rates nearing 100%. A survey of rodents captured in the village of Soromba (rural commune of Sibirila, district of Bougouni, Mali) found that 25% of Mastomys natalensis had evidence of Lassa virus infection.

The purpose of this study is to determine the proportion of people who have been previously exposed to Lassa virus, as well as the one-year incidence of infection in three villages within the rural commune of Sibirila, district of Bougouni. We will obtain 2 fingerstick blood samples (approximately one year apart) from each of approximately 600 participants aged greater than or equal to 6 months. Participants will be passively followed for one year and asked to present to their local health center if they have a fever.

Elucidation of the prevalence of Lassa virus infection in the populations living in or near Sibirila may help Malian authorities to improve surveillance and/or local diagnostics. Accurate identification of Lassa virus infections in humans will help reduce the morbidity and mortality of those living in this area.

The incidence and etiology of vector-borne diseases in southern Mali is relatively unknown. It is possible to use these samples to screen for other vector-borne diseases using similar serological assays. Expanding the testing to include filoviruses, bunyaviruses, alphaviruses and flaviviruses would greatly benefit our knowledge of circulating pathogens in southern Mali as well as the public health by helping to reduce the morbidity and mortality of those living in the area.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 6 months.
* Resident of Soromba, Bamba or Banzana with no plans to relocate within 1 year.

EXCLUSION CRITERIA:

* Any condition that in the opinion of the investigator would render the participant unable to comply with the protocol (e.g., psychiatric disease).
* Any health condition that would confound data analysis or pose unnecessary exposure risks to study personnel in the opinion of the investigator.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2014-12-05; Primary Completion 2016-10-31 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
To determine the seroprevalence of Lassa virus infection in the population of Southern Mali at the study start date. The prevalence of Lassa virus infection will be based on serological evidence in the villages of Soromba, Bamba and Banzana. | At time of study start.
To determine the proportion of individuals in these villages who haveexperienced symptoms consistent with Lassa fever at the start of the study | At time of study start.
To determine the annual incidence of seroconversion due to Lassa virus infection. Prevalence of Lassa virus exposure at the start of the study will be compared to the prevalence at the end of one calendar year to determine the one year incidence... | One year after study start date.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich U Feldmann, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Atkin S, Anaraki S, Gothard P, Walsh A, Brown D, Gopal R, Hand J, Morgan D. The first case of Lassa fever imported from Mali to the United Kingdom, February 2009. Euro Surveill. 2009 Mar 12;14(10):19145. PMID 19317988
- [Background] Safronetz D, Sogoba N, Lopez JE, Maiga O, Dahlstrom E, Zivcec M, Feldmann F, Haddock E, Fischer RJ, Anderson JM, Munster VJ, Branco L, Garry R, Porcella SF, Schwan TG, Feldmann H. Geographic distribution and genetic characterization of Lassa virus in sub-Saharan Mali. PLoS Negl Trop Dis. 2013 Dec 5;7(12):e2582. doi: 10.1371/journal.pntd.0002582. eCollection 2013. PMID 24340119
- [Background] Sogoba N, Feldmann H, Safronetz D. Lassa fever in West Africa: evidence for an expanded region of endemicity. Zoonoses Public Health. 2012 Sep;59 Suppl 2:43-7. doi: 10.1111/j.1863-2378.2012.01469.x. PMID 22958249